CLINICAL TRIAL: NCT03836638
Title: The Impact of Age on Botulinum Toxin Potency in Facial Rhytides Treatment: A Prospective Randomized Controlled Trial
Brief Title: The Impact of Age on Botulinum Toxin Potency in Facial Rhytides Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St Joseph University, Beirut, Lebanon (Other)
Responsible Party: Principal Investigator, samer jabbour, Resident, St Joseph University, Beirut, Lebanon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USJ-09
Record Dates: First submitted 2018-08-24; First posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Aging; Botulinum Toxin; Facial Wrinkles
Keywords: Botulinum Toxin; Rejuvenation; Age; Wrinkles; Rhytidis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose young subjects (Experimental): Group 1 patients will be 25-35 years old and will be injected with 30 units of botulinum toxin into the upper face
  Interventions: Drug: 30 Units of botulinum toxin
- Low dose older subjects (Experimental): Group 2 patients will be older than 45 and will be injected with 30 units of botulinum toxin into the upper face
  Interventions: Drug: 30 Units of botulinum toxin
- high dose older subjects (Active Comparator): Group 3 patients will be older than 45 and will be treated with the usual 50 units dose into the upper face (control group)
  Interventions: Drug: 50 Units of botulinum toxin

INTERVENTIONS:
Drug: 30 Units of botulinum toxin — 30 Units of botulinum toxin to upper face
  Arms: Low dose older subjects; Low dose young subjects
Drug: 50 Units of botulinum toxin — 50 Units of botulinum toxin to upper face
  Arms: high dose older subjects

SUMMARY:
Botulinum toxin is approved by the FDA for the treatment of facial wrinkles. Patients are usually older than 45 years and their main demand is to treat pre-existing facial wrinkles. However with the increasing popularity of this technique, younger patients, aged 25 to 35 years, are now seeking botulinum toxin injection as a preventive measure for rhytides. The usual dose used for the treatment of facial rhytides in a female patient older than 45 years is 50 units. No consensus exists concerning the dose of botulinum toxin that should be used in younger patients. Hypothesis: lower dose of botulinum toxin is sufficient to give good and long lasting results in young patients. The objective of this randomized open-label study is to evaluate the effect of lower doses of Botulinum toxin on the facial rythides in young patients.

DETAILED DESCRIPTION:
Botulinum toxin is approved by the FDA for the treatment of facial wrinkles. Patients are usually older than 45 years and their main demand is to treat pre-existing facial wrinkles. However with the increasing popularity of this technique, younger patients, aged 25 to 35 years, are now seeking botulinum toxin injection as a preventive measure for rhytides. The usual dose used for the treatment of facial rhytides in a female patient older than 45 years is 50 units. No consensus exists concerning the dose of botulinum toxin that should be used in younger patients. Hypothesis: lower dose of botulinum toxin is sufficient to give good and long lasting results in young patients.

The objective of this randomized open-label study is to evaluate the effect of lower doses of Botulinum toxin on the facial rythides in young patients.

In this trial, patients will be divided into 3 groups: Group 1 patients will be 25-35 years old and will be injected with 30 units of botulinum toxin into the upper face, group 2 patients will be older than 45 and will be injected with the same amount of botulinum toxin into the upper face and group 3 patients will be older than 45 and will be treated with the usual 50 units dose (control group). Patients older than 45 will be randomized between groups 2 and 3. Validated photonumeric scales will be used to evaluate the wrinkles at rest and with muscle contraction at 2, 4, 8, 12, 16, 20, 24 weeks post injection in the 3 groups. The patient satisfaction rate and the Physician global assessment will also be evaluated in the 3 groups. The scores will be determined by 3 independent blinded raters.

Hypothesis:

(1) the low dose will be sufficient to treat the group 1 patients and it will be insufficient to treat the group 2 patients. (2) The results will last longer in groups 1 and 3 patients compared to group 2 patients. (3) Group 1 patients treated with low doses of botulinum toxin will have similar results to the group 3 patients treated with the standard dose of botulinum toxin.

ELIGIBILITY:
Inclusion Criteria:

* female patients presenting to our clinic for Facial wrinkle treatment with botulinum toxin
* Must be between 25-35 years old to be included in group 1.
* Must be older than 45 to be included in groups 2 and 3.

Exclusion Criteria:

* Patients with previous periorbital/forehead surgery
* Patients who plucked the upper eyebrow margin
* Patients with eyebrow tatoos
* Patients with upper face botulinum toxin injection in the past 12 months
* Patients with resorbable upper face fillers injection in the past 12 months
* Patients with previous permanent upper face fillers injection
* Pregnant patients
* Lactating patients
* Patients with preexisting neuromuscular conditions (myasthenia gravis, Eaton Lambert syndrome)
* Patients using medication that could potentiate the effect of botulinum (ex: aminoglycoside antibiotics)
* Patients with sensitivity to botulinum toxin or human albumin

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes of scores of Validated photonumeric scales: Brow Positioning Scale at rest | 0, 2, 4, 8, 12, 16, 20, 24 weeks
  0-Youthful, refreshed look and high-arch eyebrow
  1. Medium-arch eyebrow
  2. Slight arch of the eyebrow
  3. Flat arch of the eyebrow, visibility of folds, and tired appearance
  4. Flat eyebrow with barely any arch, marked visibility of folds, and very tired appearance.
Changes of scores of Validated photonumeric scales: Forehead Lines Scale at rest | 0, 2, 4, 8, 12, 16, 20, 24 weeks
  0-None
  1. Minimal
  2. Moderate
  3. Deep
  4. Extreme
Changes of scores of Validated photonumeric scales: Forehead Lines Scale with contraction | 0, 2, 4, 8, 12, 16, 20, 24 weeks
  0-None
  1. Minimal
  2. Moderate
  3. Deep
  4. Extreme
Changes of scores of Validated photonumeric scales: Glabellar Lines Scale at rest | 0, 2, 4, 8, 12, 16, 20, 24 weeks
  0-No glabella lines
  1. Mild glabella lines
  2. Moderate glabella lines
  3. Severe glabella lines
  4. Very severe glabella lines
Changes of scores of Validated photonumeric scales: Glabellar Lines Scale with contraction | 0, 2, 4, 8, 12, 16, 20, 24 weeks
  0-No glabella lines
  1. Mild glabella lines
  2. Moderate glabella lines
  3. Severe glabella lines
  4. Very severe glabella lines
Changes of scores of Validated photonumeric scales: Crow Feet Scale at rest | 0, 2, 4, 8, 12, 16, 20, 24 weeks
  0-No wrinkles
  1. Mild wrinkles
  2. Moderate wrinkles
  3. Severe wrinkles
  4. Very severe wrinkles
Changes of scores of Validated photonumeric scales: Crow Feet Scale with contraction | 0, 2, 4, 8, 12, 16, 20, 24 weeks
  0-No wrinkles
  1. Mild wrinkles
  2. Moderate wrinkles
  3. Severe wrinkles
  4. Very severe wrinkles

SECONDARY OUTCOMES:
Investigators Global Aesthetic Improvement Scale | 0, 2, 4, 8, 12, 16, 20, 24 weeks
  1. Very Much Improved: optimal cosmetic results
  2. Much Improved: marked improvement in appearance from initial condition but not completely optimal
  3. Improved: obvious improvement in appearance from initial condition but additional treatments are advised
  4. No Change: the appearance is the same as the original condition
  5. Worse: the appearance is worse from the original condition
Patient satisfaction | 0, 2, 4, 8, 12, 16, 20, 24 weeks
  1. Very Satisfied
  2. Satisfied
  3. Dissatisfied
  4. Very Dissatisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Hotel Dieu De France, Beirut, Aschrafieh, Lebanon

IPD SHARING:
Plan to Share IPD: No